CLINICAL TRIAL: NCT04821947
Title: Effects of Rhomboid Intercostal Plane Block for Postoperative Analgesia After Thoracoscopic Surgery Compared With Local Anesthetic Infilteration: A Randomized Clinical Trial
Brief Title: Rhomboid Intercostal Plane Block vs Local Anesthetic Infilteration for Postoperative Analgesia After Thoracoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: FMASU R 34/2021
Record Dates: First submitted 2021-03-26; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIB Group (Active Comparator): Drug: Bupivacaine 0.25% patients will receive 20 ml of bupivacaine 0.25% in the rhomboid plane under rhomboid major muscle
  Interventions: Other: Rhomboid intercostal plane block or Local anesthetic infiltration of 0.25% Bupivacaine
- LA Group (Active Comparator): Drug: Bupivacaine 0.25% patients will receive wound infiltration of VATS incision, single-incision with 10mL 0.25% bupivacaine double-incision with 15 mL (10mL+5mL) 0.25% bupivacaine three-port strategy with 17 mL (10mL+5mL+2mL) 0.25% bupivacaine .
  Interventions: Other: Rhomboid intercostal plane block or Local anesthetic infiltration of 0.25% Bupivacaine

INTERVENTIONS:
Other: Rhomboid intercostal plane block or Local anesthetic infiltration of 0.25% Bupivacaine — for RIB GroupThe following structures will be identified from superficial to deep: trapezius muscle, rhomboid major muscle, intercostal muscles between ribs, pleura, and lung. The tissue plane between the rhomboid major and intercostal muscles will be identified. A 18 gauge Tuohy needle will be advanced in plane from a superomedial-to-inferolateral direction, through the trapezius and rhomboid major muscles. The skin entry point for the first injection will be the T5-T6 level just medial to the scapula.
  After the location is confirmed through hydrodissection of 3 ml on the upper intercostal muscles under the rhomboid major muscle, 20ml of bupivacaine (concentration 0.25%) is injected under rhomboid major muscle LA group will receive wound infiltration of VATS incision single-incision with 10mL 0.25% bupivacaine double-incision with 15 mL (10mL+5mL) 0.25% bupivacaine three-port strategy with 17 mL (10mL+5mL+2mL) 0.25% bupivacaine

SUMMARY:
The purpose of the study is to evaluatethe effects of rhomboid intercostal block( RIB ) on postoperative pain after thoracoscopic surgery compared with local anesthetic infiltration ( LA )

ELIGIBILITY:
Inclusion Criteria:

* ASA status I &II

Exclusion Criteria:

* Allergic constitution
* Severe cardiovascular or hepatorenal insufficiency
* Coagulation system disease
* Injection site infection
* Morbid obesity (BMI>40 kg/m2).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Total amount of postoperative analgesic consumption | First 24 hours postoperative
  total dose of postoperative tramadol and morphine
Visual Analogue Score ( VAS ) | First 24 hours postoperative
  VAS will be measured at 1st, 2nd, 4th, 6th, 12th, 24th hours postoperative at rest and during cough